CLINICAL TRIAL: NCT03456791
Title: Evaluation of Serum Human Epididymis Secretory Protein 4 (HE4) in Benign Endometrial Disease and Endometrial Cancer
Brief Title: Human Epididymis Protein 4 in Endometrial Carcinoma
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Hayam Fathy Mohammad, Assisted professor of obstetrics and gynecology, Ain Shams University
Other Study IDs: 4
Record Dates: First submitted 2018-03-01; First posted 2018-03-07 (Actual); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Endometrial Cancer
Keywords: Epididymal secretory protein E4; Major epididymis specific protein E4
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood sample for polymerase chain reaction for human epididymis protein 4. endometrial sample in formalin for pathological examination
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- endometrial carcinoma( cases): 42 patients with abnormal uterine bleeding and diagnosed endometrial cancer at prior endometrial biopsy, underwent staging laparotomy will be subjected to withdrawal of blood sample for measurement of human epididymis protein 4
  Interventions: Diagnostic Test: Human epididymis protein 4
- benign diseases(control): 42 patients with abnormal uterine bleeding and diagnosed benign endometrial pathology by endometrial biopsy will be subjected to withdrawal of blood sample for measurement of human epididymis protein 4
  Interventions: Diagnostic Test: Human epididymis protein 4

INTERVENTIONS:
Diagnostic Test: Human epididymis protein 4 — Human epididymis protein will be quantitatively assayed using the enzyme immunometric assay (EIA) method
  Other Names: Major epididymis specific protein E4; putative protease inhibitor WAP5

SUMMARY:
Endometrial cancer represents the most common gynecologic cancer, and it is expected to become an even greater public health concern as the prevalence of obesity, one of the most common risk factors for endometrial cancer, increases worldwide.

Almost 20% of patients with endometrial cancer are in the premenopausal state and 10% are asymptomatic. In such a case, it is much harder to make an early diagnosis and usually they are probably diagnosed at advanced stages.

An earlier diagnosis represents an imperative goal to improve survival and prognosis of patients of endometrial cancer. Actually, there are no certified screening tools for endometrial cancer. Pelvic ultrasound as screening for endometrial cancer-reaches 80.5% of sensitivity, when endometrial echo is > 5 mm, but it dramatically decreases to 20% in asymptomatic women; moreover, specificity is low (61%).

DETAILED DESCRIPTION:
Human epididymis protein 4, a putative protease inhibition containing two Whey Acid Protein domains, is significantly increased in the endometrioid subtype of endometrial carcinoma.

Tissue microarray and polymerase chain reaction studies confirmed a high level of human epididymis 4 expression in both endometrioid and serous types of endometrial carcinoma , these results are consistent with those from other laboratories showing increased human epididymis protein 4 messenger ribonucleic acid and protein expression in endometrial cancer tissues.

Subsequent investigation demonstrated that human epididymis protein 4 are detectable in various normal tissues with varying expression levels, yet their levels are significantly increased in endometrial carcinoma compared to normal endometrium.

Human epididymis protein 4 ( HE4) is a member of the whey-acidic protein family and it is . Human epididymis protein 4 was first isolated from the human epididymis .

This protein is also known as epididymal secretory protein E4, major epididymis specific protein E4 and putative protease inhibitor WAP5. WFDC-2 gene product was originally thought to be a protein specifically expressed in the epididymis and was dubbed as a tissue marker for the same.

Angioli etal 2013, found HE4 cutoff of 70pmol/l yields the best sensitivity and specificity for detecting endometrial cancer (59.4%) sensitivity and 100% specificity) with a positive predictive value 100% and negative predictive value equal to 71.52% for the 70 pmol/l cutoff, also found that HE4 marker was never increased in patients with benign diseases Kalogera etal 2012 found that HE4 is elevated in high proportion of endometrial cancer patients and it is correlated with myometrial invasion (> 50% P< 0.00) also found that lymph node, statue correlates with the HE4 values there is a statistical significant difference comparing stage I versus stage III (P < 0.0010).

These findings suggest that HE4 could be useful as a preoperative indicator to identify patients suitable for pelvic and para aortic lymphadenectomy.

ELIGIBILITY:
Inclusion Criteria:

* Age (45 - 70 yr old).

Exclusion Criteria:

1. Age more than 70 yr and less than 40 yr.
2. Abnormal cardiac hematological renal hepatic functions.
3. Breast cancer or other malignancies.
4. Concomitant benign and for malignant adnexal pathologies.
5. Hormonal medication.
6. Patient taking or having chemo-radiotherapy.
7. Patients unfit for surgical intervention.
8. Smoker.

Ages: 45 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: 1- History taking, general examination , pelvic ultrasound will be done for all patients under the study,endometrial biopsy will be obtained form all patients and will be reviewed by the pathologists.
  6- Computed axial tomography (CT scan) will be done for patient with endometrial carcinoma (case study) for detect tumor as a part of metastatic workup.
  7- Pre-operative complete investigation will be done for patient underwent staging lapratomy (CBC, kidney function tests , liver function tests, FBS and coagulation profile to rule out systemic causes of bleeding.
  8- Blood sample will be taken from all patients to assess serum level of HE4.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
Relation between preoperative level of human epididymis protein 4 and surgicopathological staging of endometrial carcinoma | one week
  following staging laparotomy for cases of endometrial carcinoma , the result of pathology will be correlated to HEP4

CONTACTS AND LOCATIONS:
Overall Officials: Hayam F Mohammad, MD, Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Egypt